CLINICAL TRIAL: NCT02448030
Title: Effects of Functional Electrical Stimulation Compared to Isometric Exercise on Metaboreflex Activation in Healthy Individuals: Randomized Crossover Clinical Trial
Brief Title: Effects of Functional Electrical Stimulation on Metaboreflex Activation in Healthy Individuals
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Beatriz D'Agord Schaan, Doctor, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0359
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Reduction of Blood Flow
Keywords: Metaboreflex; Variation of blood flow; Functional electrical stimulation; Isometric exercise.
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional electric stimulation (Experimental): Other: The FES will be placed at the flexor muscles of the forearm and knee extensors, for evaluation of upper and lower limbs, respectively.
  Interventions: Other: Functional electric stimulation
- Isometric exercise (Placebo Comparator): For the upper limbs the isometric contraction exercise with handgrip will be performed for 5 minutes with 30% of loading, previously measured by maximum voluntary contraction test.
  Interventions: Other: Isometric exercise

INTERVENTIONS:
Other: Functional electric stimulation — The FES will be placed at the flexor muscles of the forearm and knee extensors, for evaluation of upper and lower limbs, respectively. The stimulation frequency will be 20 Hz. The pulse width used will be 0.5 milliseconds and the contraction time will be 60 seconds (TON: 60s) with a 1-second rest interval (TOFF: 1s). The total time of application will be determined for the muscle fatigue that will be evaluated by 10-point Borg scale and by the measurement of lactate accumulation that must not exceed 30 minutes. The intensity will be adjusted individually, taking into account the patient's ability to promote the full flexion of the wrist / knee extension and comfort during contractions. Along with the application of FES a 1 Kg overload will be applied to intensify the fatigue time.
  Other Names: FES
  Arms: Functional electric stimulation
Other: Isometric exercise — For the upper limbs the isometric contraction exercise with handgrip will be performed for 5 minutes with 30% of loading, previously measured by maximum voluntary contraction test. For the lower limbs the knee extension exercise will be conducted in a training station. The SBP, DBP, MBP and HR will be recorded through the protocols. Fatigue will be determined every minute by the 10-point Borg scale and by measurement of lactate accumulation before, immediately after the protocol, and 5 minutes during the recovery period.
  Arms: Isometric exercise

SUMMARY:
Cardiovascular exercise adjustments are required during in order to redistribute blood flow from non-exercising vascular areas to active muscles. This hemodynamic adjustments, which are partially mediated by mechanosensitive and metabosensitive reflexes, ultimately increase oxygen and nutrient delivery to exercising muscle tissues (Mitchell, 1990). Static handgrip exercise has been shown to induce alterations in the arterial baroreflex function (Kim, 2005) and activation of muscle metaboreflex that increases arterial blood pressure and peripheral vasoconstriction, respectively. Functional electrical stimulation (FES) treatment used in physical therapy in patients who are unable to tolerate conventional exercise showed to be a good alternative for muscle strengthening (Sbruzzi, 2010) and to improve metabolic abnormalities (Karavidas, 2006). However, the effect of FES on metaboreflex activation in healthy individuals has never been investigated. Therefore, this study aims to evaluate the metaboreflex activation induced by FES in upper and low limbs in healthy individuals, and also to compare their results with the effects caused by isometric exercise.

DETAILED DESCRIPTION:
All participants will be invited to attend four separate days for completion of the study protocols. On the first day, the metaboreflex activation in upper limb will be randomly assigned to isometric exercise or FES intervention. On the second day, at least two days apart, random isometric exercise or FES intervention will be performed in the upper limb. On the third day, at least one week apart, all participants will be assigned to perform metaboreflex in a lower limb induced by isometric exercise or FES intervention. On the fourth day, at least two days apart, random isometric exercise or FES intervention will be performed in a lower limb. To evaluate the isometric exercise and FES intervention the post-exercise ischemia will be randomly performed to evaluate the accumulation of metabolites in response to activated limb (PECO +) and evaluation control without ischemia (PECO-). The experiments between PECO+ and PECO- will be separated by a 30 min interval. During isometric exercise and FES protocols the blood flow and peripheral vascular resistance will be assessed by venous occlusion plethysmography. Fatigue will be determined every minute by the 10-point Borg scale to assess rate of perceived exertion and by blood lactate. Blood lactate will be evaluated through capillary action at pre, immediately post exercise and at 5 minutes during the recovery period. Hemodynamic variables such as BP and HR will be recorded every minute during the protocols.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Both genders
* Aged 35-70 years
* Sedentary
* Not using continuous medications

Exclusion Criteria:

* Cardiovascular disease
* Neurological disease
* Malignant disease
* Peripheral vascular disorders (varicose veins or deep vein thrombosis)
* Peripheral sensitivity alterations
* Contraindication to performing physical exercise
* Refusal to sign the consent form

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Forearm and calf blood flow change | 5 minutes of exercise ( when PECO-) or to fatigue (when PECO +)
  When performed the protocol with FES measurements will be taken for 3 minutes of rest (in both PECO+ and PECO-), 5 minutes of exercise (when PECO-) or to fatigue (when PECO +), during the 3 minutes of occlusion (when PECO +) and 3 minutes final recovery (in both PECO+ and PECO-). When performed the protocol with isometric exercise measurements will be at 3 minutes basal (in both PECO+ and PECO-), 3 minutes of exercise (in both PECO+ and PECO-), 3 minutes of occlusion when PECO + and 3 minutes of ultimate recovery (in both PECO+ and PECO-).

SECONDARY OUTCOMES:
Maximum muscle strength | The maximum peak strength will be measured 3 times with 1 minute interval between each measurement before a session of isometric exercise
  Before starting the evaluations of blood flow, the maximum peak strength is measured three times with 1 minute interval between each measurement, after is calculated 30% of the maximum value and the determined load exercise.
Peripheral vascular resistance | It is calculated using data obtained from blood flow and mean arterial pressure in the protocols at 3 minutes in both PECO+ and PECO-
  Ratio between the mean arterial pressure (MBP) and muscle blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Dr Schaan, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre; Aline Macedo, Graduate, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Mitchell JH. J.B. Wolffe memorial lecture. Neural control of the circulation during exercise. Med Sci Sports Exerc. 1990 Apr;22(2):141-54. No abstract available. PMID 2192221
- [Background] Rowell LB, O'Leary DS. Reflex control of the circulation during exercise: chemoreflexes and mechanoreflexes. J Appl Physiol (1985). 1990 Aug;69(2):407-18. doi: 10.1152/jappl.1990.69.2.407. PMID 2228848
- [Background] Kim JK, Sala-Mercado JA, Rodriguez J, Scislo TJ, O'Leary DS. Arterial baroreflex alters strength and mechanisms of muscle metaboreflex during dynamic exercise. Am J Physiol Heart Circ Physiol. 2005 Mar;288(3):H1374-80. doi: 10.1152/ajpheart.01040.2004. Epub 2004 Nov 11. PMID 15539416
- [Background] Sbruzzi G, Ribeiro RA, Schaan BD, Signori LU, Silva AM, Irigoyen MC, Plentz RD. Functional electrical stimulation in the treatment of patients with chronic heart failure: a meta-analysis of randomized controlled trials. Eur J Cardiovasc Prev Rehabil. 2010 Jun;17(3):254-60. doi: 10.1097/HJR.0b013e328339b5a2. PMID 20560163
- [Background] Karavidas AI, Raisakis KG, Parissis JT, Tsekoura DK, Adamopoulos S, Korres DA, Farmakis D, Zacharoulis A, Fotiadis I, Matsakas E, Zacharoulis A. Functional electrical stimulation improves endothelial function and reduces peripheral immune responses in patients with chronic heart failure. Eur J Cardiovasc Prev Rehabil. 2006 Aug;13(4):592-7. doi: 10.1097/01.hjr.0000219111.02544.ff. PMID 16874150